## Pain Modulatory Profiles in Stretching NCT05891353 8/26/2024

## STUDY PROTOCOL

This study was a crossover trial of healthy participants. After providing written informed consent, participants were screened for eligibility criteria. Eligible participants then underwent three interventions across three separate sessions. First, participants completed a cold water immersion task that included immersion of the dominant hand in a bath of water for 1 minute, 4 times. Second, participants completed a pain inducing stretching in which they underwent stretching of the upper trapezius for a moderate intensity for 1 minute, 4 times. Third, participants underwent a pain free stretch in which they underwent stretching of the upper trapezius for a low intensity for 1 minute, 4 times. Between each minute, pressure pain threshold was assessed at the non-dominant webspace of the foot.

## STATISTICAL ANALYSIS

To examine the immediate changes in PPT by condition, a repeated measures ANOVA was conducted. Simple effects decomposition with Bonferroni correction were completed. Our a priori alpha level is <0.05.